CLINICAL TRIAL: NCT04430660
Title: Evaluating Glial Acetate Metabolism as a Biomarker of Hypoglycemic Complications in Diabetic Patients: A Proof of Concept Study.
Brief Title: Evaluating Glial Acetate Metabolism as a Biomarker of Hypoglycemic Complications in Diabetic Patients
Acronym: GLEAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, David McDougal, Assistant Professor, Pennington Biomedical Research Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PBRC 2018-060
Record Dates: First submitted 2020-01-16; First posted 2020-06-12 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Diabetes; Hypoglycemia
MeSH Terms: conditions — Diabetes Mellitus; Hypoglycemia | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Other): Participants will have there glial acetate metabolism assessed via 13C MRS at baseline and then again 14 days later. Participants will wear blinded continuous glucose monitoring devices for ~4 weeks.
  Interventions: Other: 13C-MRS procedure/Acetate infusion; Device: Continuous glucose monitoring

INTERVENTIONS:
Other: 13C-MRS procedure/Acetate infusion — Glial metabolism will be measured via MRS utilizing a simultaneous intravenous infusion of 13C labeled acetate. An intravenous catheter will be placed in a vein of each arm, one to infuse 13C-acetate and the other to draw blood samples.
Device: Continuous glucose monitoring — Participants will wear blinded continuous glucose monitoring devices (dexcom, G6) for approximately 4 weeks. Sensors will be replaced every 7-10 days.
  Other Names: CGM

SUMMARY:
A recent pilot study, GLIMPSE (NCT02690168), was recently completed which demonstrated that the rate of glial acetate metabolism (GAM) is closely associated with susceptibility to fasting-induced hypoglycemia in healthy adults. Insulin-induced hypoglycemia is a common complication of diabetes treatment and is a major barrier to the maintenance of healthy glucose levels in individuals with diabetes. The primary purpose of the study is to test the proof-of-concept that there is an association between the rate of GAM and susceptibility to insulin-induced hypoglycemia. In order to observe such a relationship the rate of GAM will be measured in a patient population known to frequently experience hypoglycemia, i.e., individuals with type 1 diabetes mellitus (T1DM).

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Ages 18-40 years
* Diagnosed with type 1 diabetes with positive antibodies or dependent on insulin therapy
* HbA1c of ≤8.5%
* Modified Clarke's Hypoglycemia Questionnaire score of 12-24
* Willing to participate in continuous glucose monitoring (CGM)

Exclusion Criteria:

* Contraindication to MRI
* Consume >10 alcoholic drinks/week
* Current use of CGM
* Current use of insulin pump
* Current use of any diabetes medication other than insulin, e.g. SGLT1/2 inhibitors.
* Current use of steroids, e.g. cortisone, and prednisone.
* History of chronic smoking or have quit less than 10 years ago
* History of cancer in the past 5 years (individuals with basal cell or squamous cell skin cancer would be allowed)
* History of seizures
* Significant, cardiac, vascular, pulmonary, gastrointestinal, neurologic, hematologic, rheumatologic, or psychiatric disease
* Significant liver disease as defined as more than twice the upper limit of normal for liver enzymes
* Significant renal disease as defined as a estimated glomerular filtration rate less than 30
* Pregnant, planning to become pregnant, or breastfeeding
* Have been hospitalized or treated in the past 3 months for severe hypoglycemia
* Based on the investigative team's clinical judgement, a subject may not be appropriate for participation in the study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2020-08-19 (Actual); Primary Completion 2022-03-29 (Actual); Study Completion 2022-05-04 (Actual)

PRIMARY OUTCOMES:
Change in percent 13C enrichment of bicarbonate measured via carbon-13 magnetic resonance spectroscopy (13C-MRS) | Once at Study Visit 1 day and 1 day at Study Visit 3, 14 days apart

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana
  - Tulane Medical Center, New Orleans, Louisiana